CLINICAL TRIAL: NCT00133159
Title: A Double-Blind Phase IIb Study to Evaluate the Safety and Efficacy of Different Doses of Tyrosine Adsorbed Grass/Rye Pollen Allergoid With MPL in Patients Sensitized to Grass and Rye Pollen
Brief Title: Different Doses of Tyrosine Adsorbed Grass Pollen Allergoid With Monophosphoryl Lipid A (MPL) in Patients Sensitized to Grass Pollen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergy Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GrassMATAMPL203; P2DP5005
Record Dates: First submitted 2005-08-22; First posted 2005-08-23 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Type I Hypersensitivity
Keywords: Allergy; Specific Immunotherapy
MeSH Terms: conditions — Hypersensitivity, Immediate; Hypersensitivity

INTERVENTIONS:
Biological: Grass MATAMPL

SUMMARY:
Allergen-specific immunotherapy (SIT), the administration of gradually increasing quantities of an allergen extract to an allergic patient, is a curative approach which directly treats the underlying allergic disease. GrassMATAMPL has been developed to provide pre-seasonal specific immunotherapy for patients with an allergy to grass pollen (hay fever). The purpose of this double-blind Phase IIb study is to assess the tolerability and immunogenicity of different doses of GrassMATAMPL in volunteers allergic to grasses and rye pollen.

ELIGIBILITY:
Inclusion Criteria:

* positive skin prick test for grass and rye allergen
* Specific IgE for grass and rye as documented by radioallergosorbent or equivalent test with class >= 2
* History of at least 1 season of moderate to severe seasonal rhinoconjunctivitis due to an IgE - mediated allergy to pollen from grass and rye
* Males or non-pregnant, non-lactating females who are post-menopausal or naturally or surgically sterile. Females of childbearing potential have a confirmed absence of pregnancy according to a negative urine pregnancy test and must be using an acceptable birth control method.
* Spirometry at Screening demonstrates FEV1 >= 80% predicted and FEV1/FVC >= 70%

Exclusion Criteria:

* Acute or subacute atopic dermatitis and/or urticaria factitia and/or urticaria due to physical or chemical influence and/or chronic dermatitis
* Patient has moderate to severe asthma
* Visual inspection of the forearms indicates potential problems with the conduct or interpretation of the skin prick test; both forearms must be available for testing
* History or presence of diabetes, cancer or any clinically significant cardiac, metabolic renal, hematologic diseases or disorders
* Recent clinically significant history (within 2 years) of hepatic gastrointestinal, dermatologic, venereal, neurologic or psychiatric diseases or disorders
* Any clinically significant (as determined by the investigator) abnormal laboratory value
* Perennial allergens: clinically relevant sensitivity against house dust mites, molds, and epithelia
* Patient has clinically relevant sensitivity against the following summer/autumn season flowering plants: plantain, orache, nettle, mugwort, Bermuda grass, or ragweed.
* Secondary alteration at the affected organ
* History of autoimmune diseases and/or rheumatoid diseases
* Patient is taking b-blockers
* Patient who is not allowed to receive adrenalin
* Patients in whom tyrosine metabolism is disturbed
* Presence of a disease with a pathogenesis interfering with the immune response and patient has received medication which could influence the results of this study
* Documented evidence of acute or significant chronic infection
* History of anaphylaxis
* Documented history of angioedema
* Hypersensitivity to excipients in the study medications
* Previous or current immunotherapy with comparable grass/rye allergen extracts
* Currently using anti-allergy medication and other drugs with antihistaminic activity
* Patients currently participating in a clinical trial or who have been exposed to study medication within the last 30 days
* Patient is pregnant or planning pregnancy and/or lactating
* Patient has received treatment with preparation containing MPL® during the past 12 months
* Any systemic disorder that could interfere with the evaluation of the study medication(s)
* Clinical history of drug or alcohol abuse that would interfere with the patient's participation in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68
Dates: Start 2005-09-12 (Actual); Primary Completion 2005-11-08 (Actual); Study Completion 2005-11-08 (Actual)

PRIMARY OUTCOMES:
immunological response to the three GrassMATAMPL treatment arms compared to placebo (grass specific)

SECONDARY OUTCOMES:
tolerability of different subcutaneous doses
tolerability of the cumulative subcutaneous doses
clinical chemistry and hematology
number of adverse events
number of adverse reactions
immunological response to the three GrassMATAMPL treatment arms compared to placebo (rye specific)

CONTACTS AND LOCATIONS:
Overall Officials: Kemi Oluwayi, MD, Study Chair — Allergy Therapeutics
Locations (3):
- Canada (3):
  - Allied Research International Inc., Mississauga, Ontario
  - Mississauga, Ontario
  - Ottawa Allergy Research Corporation, Ottawa, Ontario